CLINICAL TRIAL: NCT05134753
Title: Platelet Rich Fibrin Versus Advanced Platelet Rich Fibrin as Bone Graft Material in Sinus Augmentation (Randomized Controlled Clinical Trial)
Brief Title: PRF Versus Advanced PRF in Sinus Augmentation
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mahinour magdy mohamed, Resident oral surgery, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: PRF and sinus augmentation
Record Dates: First submitted 2021-11-15; First posted 2021-11-26 (Actual); Last update posted 2021-12-23 (Actual); Status verified 2021-12

CONDITIONS: Maxillary Sinus
Keywords: PRF; Advanced PRF; Sinus augmentation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study arm (Experimental): Patients will undergo sinus augmentation with advanced PRF
  Interventions: Biological: Advanced PRF
- Controlled arm (Placebo Comparator): Patients will undergo sinus augmentation with PRF
  Interventions: Biological: Control

INTERVENTIONS:
Biological: Advanced PRF — Advanced PRF will be placed for patients undergoing sinus augmentation
  Arms: Study arm
Biological: Control — PRF will be placed for patients undergoing sinus augmentation
  Arms: Controlled arm

SUMMARY:
In the present study the main hypothesis , Advanced PRF will improve the bone quality and quantity in sinus augmentation

ELIGIBILITY:
Inclusion Criteria:

* The Patients with missing posterior maxillary teeth with insufficient available bone for implant placement indicating the need for maxillary sinus floor augmentation before implantation.

  2. The Patients should be free from any systemic disease that may affect normal healing of bone, and predictable outcome.

  3. The Patients should be free from any sinus disease that might affect the health and integrity of the sinus lining.

  4. Assign an informed consent to be involved in the study.

Exclusion Criteria:

Patients with any systemic disease that may affect normal healing. 2. Patients with any sinus disease.

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-01-30 (Estimated); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Bone quality | Six months
  Histological analysis for core biopsies Available bone quality will be evaluated by measuring the Total Bone Volume (TBV)

SECONDARY OUTCOMES:
Bone quantity | Six months
  • Linear height measurements changes of the bone will be evaluated via panoramic X-rays

IPD SHARING:
Plan to Share IPD: No